CLINICAL TRIAL: NCT03592511
Title: Effect of the Consumption of Burgers Prepared With Wine Grape Pomace Flour, Rich in Fiber and Antioxidants, on Components of the Metabolic Syndrome in Humans
Brief Title: Effect of the Consumption of Burgers Prepared With Wine Grape Pomace Flour, on Components of the Metabolic Syndrome
Acronym: WGPF-burger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Inés Urquiaga, Associate investigator, Pontificia Universidad Catolica de Chile
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15-122; IT14I10011 (Other Grant/Funding Number: FONDEF)
Record Dates: First submitted 2018-06-21; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Food Selection; Metabolic Syndrome
Keywords: Intervention study; Functional food; Grape pomace
MeSH Terms: conditions — Food Preferences; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): WGPF-burger group
  Interventions: Dietary Supplement: WGPF-burger; Dietary Supplement: Control-burger
- Control (Placebo Comparator): Control-burger group
  Interventions: Dietary Supplement: Control-burger

INTERVENTIONS:
Dietary Supplement: WGPF-burger — Volunteers consumed a WGPF-burger daily
  Arms: Intervention
Dietary Supplement: Control-burger — Volunteers consumed a Control-burger daily

SUMMARY:
Wine grape pomace flour (WGPF) is a fruit byproduct high in fiber and antioxidants. The effect of WGPF consumption was tested on blood biochemical parameters including oxidative stress biomarkers. In a 3-month intervention study, 27 male volunteers, each with some components of metabolic syndrome, consumed a beef burger supplemented with 7% WGPF containing 3.5% of fiber and 1.2 mg GE/g of polyphenols (WGPF-burger), daily during the first month. The volunteers consumed no burgers in the second month, and one control burger daily in the third month. At baseline and after these periods, there were evaluated metabolic syndrome components, plasma antioxidant status [2,2-diphenyl-1-picrylhydrazyl radical scavenging capacity (DPPH),uric acid, vitamin E, vitamin C], and oxidative damage markers [advanced oxidation protein products (AOPP), oxidized low-density lipoproteins (oxLDL), malondialdehyde (MDA)].

DETAILED DESCRIPTION:
The intervention was carried out at workplaces in Santiago, Chile. Workers were informed about the study and invited to participate. Initially, 34 male workers meeting all criteria agreed to partake, however 27 workers completed the study. Seven volunteers quit the study because three disliked the blood sampling procedure, two were sent to work abroad, one left the workplace, and one presented gastrointestinal symptoms associated with WGPF-burger consumption.

The volunteers entered a longitudinal trial consisting of two treatment periods of 4 weeks, separated by a third four-week wash-out period. For the first 4 weeks, they consumed one WGPF-burger daily, then they were washed-out and finally they consumed one control-burger daily during 4 weeks. They were asked to maintain their regular eating habits and lifestyle during the study, except for the daily intake of burgers during the treatment periods. The burgers were eaten in replacement of red or processed meat consumption, or in addition to their regular meal when it did not contain meat products. During the washout period, all subjects consumed their usual diet. Burger intake was supervised every day at lunch at the canteens of the workplaces. On weekends, participants were asked to consume burgers at home with their regular meals. In addition, compliance with burger consumption was carefully monitored by frequent calls from the dietitian.

Blood samples were obtained at weeks 0, 4, 8, and 12 for analysis. Participants had clinical, nutritional, and anthropometric evaluations at the beginning and the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were having at least one of the five components of metabolic syndrome and a BMI between 25.0 and 39.9 kg/m2

Exclusion Criteria:

* Exclusion criteria were use of drug therapy for diabetes mellitus, hypertension, or dyslipidemia and intake of pharmacological treatment with drugs that modify plasma antioxidant capacity or inflammation.

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2016-10-15 (Actual); Study Completion 2016-10-15 (Actual)

PRIMARY OUTCOMES:
Metabolic syndrome components | Month 1, WFPG-burger consumption
  The presence of metabolic syndrome components was defined using the criteria proposed by the Adult Treatment Panel III of the US National Cholesterol Education Program: (i) abdominal obesity as waist circumference >102 cm for men; (ii) low levels (<40 mg/dL for men) of serum high density lipoprotein cholesterol; (iii) hypertriglyceridemia as 150 mg/dL or more; (iv) elevated blood pressure as 130/85 mm Hg or higher; and (v) impaired glucose homeostasis as fasting plasma glucose levels of 100 mg/dL or higher
Metabolic syndrome components | Month 3, control burger consumption
  The presence of metabolic syndrome components was defined using the criteria proposed by the Adult Treatment Panel III of the US National Cholesterol Education Program: (i) abdominal obesity as waist circumference >102 cm for men; (ii) low levels (<40 mg/dL for men) of serum high density lipoprotein cholesterol; (iii) hypertriglyceridemia as 150 mg/dL or more; (iv) elevated blood pressure as 130/85 mm Hg or higher; and (v) impaired glucose homeostasis as fasting plasma glucose levels of 100 mg/dL or higher

SECONDARY OUTCOMES:
Insulin | Month 1, WFPG-burger consumption
  Fasting plasma Insulin was measured by electrochemiluminescence immunoassay (ECLIA; Roche Diagnostics®).
Insulin | Month 3, control burger consumption
  Fasting plasma Insulin was measured by electrochemiluminescence immunoassay (ECLIA; Roche Diagnostics®).
Antioxidants | Month 1, WFPG-burger consumption
  Antioxidants measurements: 2,2-diphenyl-1-picrylhydrazyl radical scavenging capacity (DPPH), uric acid, vitamin E, vitamin C
Antioxidants | Month 3, control burger consumption
  Antioxidants measurements: 2,2-diphenyl-1-picrylhydrazyl radical scavenging capacity (DPPH), uric acid, vitamin E, vitamin C
Oxidative stress | Month 1, WFPG-burger consumption
  Oxidative stress markers: Advanced oxidation protein products (AOPP), oxidized low-density lipoproteins (oxLDL), malondialdehyde (MDA)
Oxidative stress | Month 3, control burger consumption
  Oxidative stress markers: Advanced oxidation protein products (AOPP), oxidized low-density lipoproteins (oxLDL), malondialdehyde (MDA)

IPD SHARING:
Plan to Share IPD: No